CLINICAL TRIAL: NCT00523588
Title: Single Blind, Controlled, Single-Center Study of Laser Treatment in Cutaneous Lupus Erythematosus
Brief Title: Treatment of Cutaneous Lupus Erythematosus (CLE) With the 595 nm Flashlamp Pulsed Dye Laser
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Dr. Victoria Werth/Professor of Medicine and Dermatology, University of Pennsylvania School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 805209
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2010-01

CONDITIONS: Cutaneous Lupus Erythematosus
Keywords: Cutaneous lupus erythematosus; Pulsed dye laser
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: laser treatment (Candela Vbeam Perfecta™) — This laser has an adjustable pulse duration (0.45-40 ms), fixed wavelength 595 nm, spot size (3 mm, 5 mm, 7 mm, and 10 mm), and incident fluence range of 10-40 J/cm2. The laser is also equipped with a dynamic cooling device (DCD) (FDA cleared under K001589) that delivers cryogen (R-134a) from a small nozzle positioned 4 cm above the skin at an angle of approximately 70 degrees with respect to the skin surface. All patients will be treated with the laser device on which the varying cooling device parameters will be selected based on the clinical judgment of the treating physician. Factors used in this decision include patient age, skin type and epidermal pigmentation, size and depth of vessels, color of lesions, anatomic location, etc. In all instances, a test-dose in an inconspicuous location on the skin will be conducted prior to the first treatment.

SUMMARY:
The purpose of using the 595 nm Vbeam Perfecta™ flashlamp-excited, pulsed dye laser in this study is to help improve study patients' skin disease. Cutaneous lupus erythematosus (CLE) often presents with disfiguring vascular lesions which are frequently difficult to treat with the available therapeutic measures, such as photoprotection, topical steroids, and antimalarials. Laser therapy provides an alternative treatment option for CLE patients. Although there has been documented experience with laser treatment in CLE patients, no study comparing treated lesions to the natural course of the disease has been conducted.

DETAILED DESCRIPTION:
The Candela Vbeam PerfectaTM is an FDA approved 595nm Flashlamp Pulsed Dye Laser (PDL) that is being used for the treatment of benign skin lesions. The purpose of using the PDL in this study is to help improve study patients' skin disease. Cutaneous Lupus Erythematosus often starts with damaging skin lesions which are frequently difficult to treat with the available therapeutic measures. This study will use a flashlamp PDL to compare treated cutaneous lesions and non-treated lesions. We will look at factors such as the degree of erythema (redness of the skin), scale and hypertrophy (increase in size of skin), scarring and dyspigmentation (abnormality in the formation or distribution of skin coloration) and make a summary score of these factors.

It is important to note that this device currently is being used to treat patients with skin lesions in the Department of Dermatology at the University of Pennsylvania, where this study will be done. Although the PDL has been used to treat other patients, its use in this study is experimental.

The PDL is considered to be the laser of choice for vascular lesions, because at wavelengths of 585-595 nm, the laser is known to produce excellent clinical results at minimal risk to patients. The laser has been used successfully in the treatment of port-wine stains in children as young as 1 month of age. The PDL is designed to deliver an intense but gentle burst of laser light to the skin. The light is absorbed by the blood vessels in the vascular lesion, while leaving the surrounding tissue undamaged. The PDL has been used clinically for the treatment of cutaneous lesions in childhood port-wine stains, childhood proliferative angiomas, facial telangiectasias, poikiloderma of Civatte, nevus flammeus, capillary hemangiomas, scars, verrucae, and lupus erythematosus. Several studies are known to have used the 585-595nm PDL to treat cutaneous lupus erythematosus lesions.

During a period of 5 months, study patients will receive 3-5 treatments to one skin lesion with the pulsed dye laser. Clinical follow-up examinations include photographs, clinical assessments by a blinded physician, and pain and itch scales by the study patient. The study requires a total of one year commitment per study patient.

ELIGIBILITY:
Inclusion Criteria:

* Cutaneous lupus erythematosus confirmed by histological analysis
* Fitzpatrick I-III skin type (very fair, fair, or medium skin)
* Stable disease and in relatively good health
* Presence of two skin lesions that are suitable for laser treatment
* Written informed consent available prior to any screening procedures
* Female patients must be willing to use the appropriate birth control measures that will prevent pregnancy from the time of signing informed consent through 60 days after their last laser treatment

Exclusion Criteria:

* Clinically significant dyspigmentation
* History of isotretinoin use, phenol peels, filler injections (collagen, fat), dermabrasion within the past 3 years
* History of hypertrophic scarring
* History of photosensitivity in the 585-600 nm wavelength region
* History of seizure disorders triggered by light
* Pregnancy and lactation
* Fitzpatrick V or VI skin type (moderately pigmented brown, or markedly pigmented black skin)
* Patients receiving anticoagulants and/or medication for which sunlight exposure is a contraindication
* Known malignancy or prior malignancy, other than non-melanoma skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-02 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Comparison of laser treated CLE skin lesions with a non-treated control CLE lesion of the same patient evaluated by the CLASI (Cutaneous Lupus Erythematosus Disease Area and Severity Index) and the M-CLASI (Modified CLASI). | One year

SECONDARY OUTCOMES:
Pain and itch relief compared to baseline and between the treated and untreated lesion | One Year
Reduction or increase in CLASI and MCLASI scores compared to baseline, and adverse events | One year

CONTACTS AND LOCATIONS:
Overall Officials: Victoria P Werth, M.D., Principal Investigator — University of Pennsylvania, Department of Dermatology and Internal Medicine
Locations (1):
- University of Pennsylvania, Department of Dermatology, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Nunez M, Boixeda P, Miralles ES, de Misa RF, Ledo A. Pulsed dye laser treatment of telangiectatic chronic erythema of cutaneous lupus erythematosus. Arch Dermatol. 1996 Mar;132(3):354-5. No abstract available. PMID 8607651
- [Background] Raulin C, Schmidt C, Hellwig S. Cutaneous lupus erythematosus-treatment with pulsed dye laser. Br J Dermatol. 1999 Dec;141(6):1046-50. doi: 10.1046/j.1365-2133.1999.03203.x. PMID 10606850
- [Background] Baniandres O, Boixeda P, Belmar P, Perez A. Treatment of lupus erythematosus with pulsed dye laser. Lasers Surg Med. 2003;32(4):327-30. doi: 10.1002/lsm.10169. PMID 12696102